CLINICAL TRIAL: NCT01775969
Title: Effect of Modality on Discharge Instruction in Patients Receiving Outpatient Antibiotic Prescriptions From the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 11-3329
Record Dates: First submitted 2013-01-23; First posted 2013-01-25 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Modality of Discharge Instructions

ARMS (3):
- Standard of Care (No Intervention): Written discharge instructions only
- Text Message (Experimental): Written discharge instructions plus a text message with antibiotic prescription instructions
  Interventions: Other: Text Message
- Voicemail (Experimental): Written discharge instructions plus a voicemail with antibiotic prescription instructions
  Interventions: Other: Voicemail

INTERVENTIONS:
Other: Text Message — A text message with instructions is sent to the patient
  Arms: Text Message
Other: Voicemail — A voicemail with instructions is sent to the patient
  Arms: Voicemail

SUMMARY:
Outpatient antibiotics are frequently prescribed from the emergency department, and limited health literacy may impact compliance with recommended treatments. The investigators are looking to determine if patient preference for multimodality discharge instructions for outpatient antibiotic therapy varies by health literacy level, and if modality effected patient-reported antibiotic compliance and 72-hour antibiotic pick-up.

DETAILED DESCRIPTION:
This is a prospective randomized trial that includes consenting patients discharged with outpatient antibiotics. Health literacy is assessed using a validated health literacy assessment, the Newest Vital Sign (NVS). Patients are randomized to a discharge instruction modality: 1) standard of care, typed and verbal medication and case-specific instructions; 2) standard of care plus text messaged instructions sent to the patient's cell phone; or 3) standard of care plus voicemailed instructions sent to the patient's cell phone. Antibiotic pick-up is verified with the patient's pharmacy at 72 hours. Patients are called at 30 days to determine antibiotic compliance.

ELIGIBILITY:
Inclusion Criteria:

* Emergency department patient being prescribed an outpatient antibiotic or the parent of a patient under the age of 18 being prescribed on outpatient antibiotic

Exclusion Criteria:

* Doesn't have a cell phone that can receive text messages and voicemail messages
* Unable to provide informed consent
* Prisoners

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2874 (Actual)
Dates: Start 2011-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
72-hour antibiotic pickup | 72 hours
  Whether or not the patient picked up their antibiotic prescription at the pharmacy
Antibiotic compliance | 30 days
  If the patient completed the entire course of antibiotics

CONTACTS AND LOCATIONS:
Overall Officials: James R Miner, MD, Principal Investigator — Hennepin Healthcare Research Institute
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States